Title: Tear Based Breast Cancer Detection

**Principal Investigator**: V. Suzanne Klimberg MD. PH.D.

Funding Sponsor: Namida Lab, Inc.

Version: 2

**Date**: 4/13/2021

# 1. Introduction and Purpose:

Namida Lab, Inc. is a biotechnology company located in Fayetteville, AR, with a certified high-complexity CLIA lab. In January of 2021, Namida Lab, Inc. completed Melody® analytical and clinical validation, a screening test for breast cancer based on proteins from tears. The validation process was carried out manually and now needs to be conducted on the Hamilton StarPlus automated ELISA system. To do this, Namida Lab, Inc. needs fifty tear samples collected from women recently diagnosed with breast cancer but who have not undergone any treatment.

# 2. Background:

## What is the Problem?

Most women recognize screening mammography as the current gold standard in breast cancer screening. However, disparities are present, leaving groups of women without adequate access to screening. Gaps in access to screening exist due to geographic location, socio-economic status, race, and ethnicity (references). In addition, studies show women who have received a false-positive result are more likely to lose trust in the current breast health continuum of care. Therefore less likely to return for follow-up screening.

### How can Melody® help?

Currently, Melody® is not intended to be a replacement for screening mammograms but an additional tool to facilitate discussion between providers and patients. Tear sample collection can be done during any routine office visit and does not require specially trained personnel. The simple collection process allows patients to be tested in a clinic they are already familiar with by personnel they already know and trust. Melody® early iteration goals are one additional piece of information gathered. One more conversation about breast health may be the key to increasing participation in annual or biennial screening mammograms.

#### Key terms

- The Clinical Laboratory Improvement Amendment (CLIA) passed in 1988 was established to provide quality standards, strengthen Federal oversight of clinical laboratories, and ensure the reliability and accuracy of patient test results. This program allows clinical labs to develop and validate the testing protocols, which can only be run in the lab where the protocol was validated.
- Namida Lab, Inc. is a CLIA certified high complexity lab.
- The FDA is responsible for developing and assigning CLIA test complexity categorization rules and guidance.
- Melody® is a high complexity lab-developed test that has been developed and validated by Namida Lab, Inc. and will be run only by Namida Lab, Inc.
- A clinical utility study evaluates the usefulness, benefits, and drawbacks of an intervention (Smart, 2006).

#### What is the Validation process for an LDT?

CLIA clearly outlines requirements for validation of a lab-developed test. In short, each assay must meet guidelines for precision, accuracy, sensitivity and specificity (both analytical and clinical), linearity and assay range. Each laboratory drafts an umbrella standard operating procedure (SOP) to conduct validation

of new assays. This SOP is then customized to each specific test the lab intends to offer. The medical director must approve all SOPs and subsequent changes to SOPs in the CLIA lab.

After completion of validation experimentation, all results are compiled in a validation report and then reviewed and approved by the medical director. All CLIA labs are under the jurisdiction of their respective state CLIA licensing boards and undergo an inspection every two years. At the time of inspection, the lab must provide validation reports for all assays available on the testing menu for review.

# What was the outcome for the validation of Melody®?

Designing the validation of Melody® was unique because there are no lab developed tests using protein biomarkers in tears to Namida Lab, Inc.'s knowledge. The nature of the sample alone provided a new level of challenge that made the validation process more stringent. Both analytical and clinical validation of Melody® was completed in January 2021. A summary of parameters analyzed and the results for the validation can be found in tables 1-2. All performance criteria were successfully achieved, and clinical validation resulted in a sensitivity of 92% and a specificity of 54%. These values were in line with previously observed sensitivity and specificity values from development work.

Table 1: Summary of Analytical Validation

| | Sample Description (Name, | | Comparison to<br>Acceptance Criteria |
|---|---|---|---|
| Study Parameter | Number, Replicates) | Results | (Pass/Fail) |
| | | Percent recovery between 80- | |
| Accuracy | 20 spiked LGF samples | 120% for all samples | Pass |
| | 24 replicates of 3 concentrations | | |
| Intra-Assay Precision | per analyte | All %CV less than or equal to 15% | Pass |
| | Duplicates of 3 concentrations | | |
| Inter-Assay Precision | 1xday for 5 days. | All %CV less than or equal to 15% | Pass |
| | | S100A8 11% 21.10 pg/ml S100A9 | |
| Sensitivity | 20 replicates of blank per protein | 14% CV 24.32 pg/ml | Pass |
| _ | | Percent difference less than 15% | |
| Linearity | 7 unknown concentrations | for all samples | Pass |

Table 2: Summary of Clinical Validation

| Study Parameter | Sample Description (Name, Number,<br>Replicates) | Results | Comparison to Acceptance<br>Criteria (Pass/Fail) |
|---|---|---|---|
| • | ' ' | | |
| Accuracy | 26 samples 3 replicates each sample | 92% | Pass |
| Sensitivity | 52 LGF samples in duplicate | 92% | Pass |
| Specificity | 50 LGF samples in duplicate | 54% | Pass |
| Stability of LGF samples | 1 pooled disease LGS | N/A | Refer to Deviations and |
| | 1 pooled non-disease LGS | | Section B, Number 4 |

# 3. Concise Summary of Project:

What exactly is Melody®?

Part 1: Tear sample collection

Tear samples are collected using a Schirmer strip, a class I medical device, typically used to test for dry eye. The filter paper strips have been repurposed to collect proteins from the ocular cavity following protocols outlined in the literature (references).

Tear collection is conducted through the following steps (figure 1):

- 1. The strip is placed in the participants' lower eyelid, and having a foreign object in the eye will cause the eye to water. The fluid released washes the inner surface of the eyelid and the ocular lens itself, allowing proteins to adhere to the strip.
- 2. The strip is left until the liquid reaches the 25 mm mark or 5 minutes has passed.
- 3. The strip is then placed in a tube containing a buffered solution and is shipped overnight to Namida Lab, Inc.



Figure 1: Collection of tear samples.

# Part 2: Clinical Lab assay

During shipment, the proteins leave the strip and go into the solution in the tube. It is this solution that is evaluated using standard ELISA techniques in the high-complexity CLIA lab. Namida Lab, Inc. is outfitted with a Hamilton Star Plus automated ELISA system. The data generated from the ELISA assay is used together with demographic information to generate a Melody® score. The score is then compared to the diagnostic threshold, and classification of High and Low will be reported.

A reference range has been developed using the distribution of Melody® scores from the clinical studies previously conducted (figure 2). In the future, this scale will be further optimized and provided to clinicians to guide their breast health discussions with patients.



Figure 2: The Melody® scale was generated using 705 samples evaluated during development and validation. Percentages in each range show the distribution of normal and breast cancer patients that fall within each range.

With validation manually completed, Namida Lab, Inc. needs to do an equivalency study on the automated robot to demonstrate consistency between manual and automated results. This analysis will

be carried out using an equal number of samples. The samples are collected from normal (i.e., recent mammogram came back with no new findings) and recently diagnosed breast cancer patients.

Namida Lab, Inc.'s Clinical Laboratory Supervisor has defined qualification criteria of 100% agreement between manual and automated validation for the validation to be considered successful.

# 4. Study Procedures:

Fifty participants will be enrolled following the timeline in Table 3. The participation is limited to a one-time sample collection.

Table 3: Study Timeline

| Objective | Wk1 Wk2 | Wk3 | Wk4 | Wk 5 | Wk6 | Wk7 | Wk8 | Wk9 | Wk 10 | Wk 11 | Wk 12 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Namida Lab clinical team to train UTMB clinic | | | | | | | | | | | |
| staff on tear collection procedures. | | | | | | | | | | | |
| Begin Study enrollment and sample acquisition | | | | | | | | | | | |
| Conduct study enrollment and sample acquisition | | | | | | | | | | | |
| Enroll last patient | | | | | | | | | | | |
| Finalize any outstanding clinical forms | | | | | | | | | | | |
| Close study | | | | | | | | | | | |

i. Data acquisition: Each participant will be provided with a questionnaire to be filled out at the time of sample collection. The study team will assist participants in answering questions such as type of breast cancer, staging information, and tumor size. If known at the time of sample collection or after the biopsy results are received. In addition, a clinical questionnaire will be filled out for each participant with specific information relating to their breast health and current diagnosis.

ii. Clinic: Visit #1

- Participant is seen
- Study eligibility is assessed
- Informed consent process
- Registration
- Questionnaires completion
- Tear sample collection

The tear sample, study participant questionnaire, and clinical info questionnaire will be shipped overnight to Namida Lab, Inc.

# 5. Sub-Study Procedures:

N/A

# 6. Criteria for Inclusion of Subjects:

Subjects may be invited to participate in this study if the individual is an adult woman and has recently been diagnosed with breast cancer.

# 7. Criteria for Exclusion of Subjects:

Subjects must be excluded from this study if they have already started treatment for the breast cancer diagnosis.

Age less than 18 or more than 100 years.

#### 8. Sources of Research Material:

Enrolled participants will be asked to complete a brief questionnaire with questions around reproductive health, personal history of cancer, and family history of cancer. In addition, a clinical questionnaire will be filled out for each participant with specific information relating to their breast health and current diagnosis. Both questionnaires can be found in the appendix section of this document.

Tear specimens will be collected from each participant.

# 9. Recruitment Methods and Consenting Process:

Potential participants will be recruited from the patient population of the study's principal investigator (PI). Suppose there are potential study participants who are not patients of the principal investigator. In that case, the potential participant will not be contacted by the study staff. Unless the potential participant has been informed of the study by their medical provider, has expressed interest in receiving more information, and/or enrolling in the study.

Individuals will be informed of the study and the opportunity to participate after diagnosis and before any treatment(s). Potential participants will be provided the information about the study, given time to review the informed consent form (IFC) and ask any questions before signing.

#### 10. Potential Risks:

Possible risks from the collection of tears are rare but include conjunctivitis or scleral or corneal abrasion. There are no known occurrences of any of these risks from the previous IRB-approved study. Any time information is collected, there is a potential risk for loss of confidentiality. Every effort will be made to keep the information confidential; however, this cannot be guaranteed.

#### 11. Subject Safety and Data Monitoring:

The Principal Investigator will monitor this study.

Due to the minimal risk to the participants and short duration of participation, this study will be reviewed on an as necessary basis from the time the IRB approves it. Suppose abnormal values are found or the testing fails in some manner. In that case, all investigators and collaborators will be informed immediately, and enrollment halted until the matter can be resolved. The patients will not be informed of their results, and the tests will not be used to decide their treatment in any way. Any unexpected or adverse events that occur, the information on events will be sent to the IRB within 30 working days.

#### 12. Procedures to Maintain confidentiality:

After sample collection, the sample will be placed in a tube with a three-to-four-digit code generated by Namida Lab, Inc. (For example, ADX-001). Corresponding labels will be provided for the study participant questionnaire, informed consent, and HIPPA form to ensure the sample and paperwork can be matched.

Completed paperwork will remain locked in the Namida Lab, Inc. facility. It will only be accessible by the clinical study staff at Namida Lab, Inc.

Any information obtained in this study will be kept confidential. Representatives from the UTMB Institutional Review Board, the United States Food and Drug Administration (FDA), or other institutional oversight offices may review records at any time. If the results of this study are published in medical literature, participant's names will not be identified.

#### 13. Potential Benefits:

Each study participant will receive a \$25.00 gift card provided by Namida Lab, Inc. for participation.

The results of the tear evaluation will not be disclosed to the patient or be used for their medical assessment or treatment.

#### 14. Biostatistics:

Clinical acceptance criteria are defined as 100% agreement between the manual and automated classification of each sample.

Namida Lab, Inc.'s CLIA Lab Medical Director established the sample size.

# 15. Appendix

# **Tear Based Breast Cancer Detection Participant Questionnaire**

# Sample ID:

Thank you for taking the time to participate in our study. Please answer the following questions to the best of your knowledge.

| Initials: | |
|---|---|
| Age: | Sex: Male Female |
| Height | Weight |
| Race: African/African American Arab/Persian Asian East Indian Hispanic/Latina | Native American White/Caucasian Multiracial Prefer not to answer |

# Section 1: In section 1 we need you to answer a few questions about your eye health:

| 1. | Have you been diagnosed <u>by a physician</u> with any of the following ocular disorders? |
|---|---|
| | Macular Degeneration |
| | Cataracts |
| | Dry Eye |
| | None |
| 2. | Have you had Lasik surgery? Yes No |
| 3. | Are you currently wearing contact lenses? No Yes right eye only left eye only |
| 4. | Have you used of the following types of eye drops today? Red eye reducing OTC for allergies |
| | Prescription steroid for allergies |
| | General hydration |
| | Saline |
| | Drops for Glaucoma |
| | Other (Please describe): |
| | None |
| | Section 2: In section 2 we will cover a few questions about your reproductive health: |
| We are | e asking the next few questions to gather information about additional hormones that you may be |
| taking. | |
| 5. | |
| | Pill Name if known: |
| | ∐Implant |
| | Contraception Injection |
| | Contraceptive Patch |
| | Intrauterine device (IUD) |
| | □ Vaginal Ring |
| | None |
| 6. | Are you currently using any type of Hormone replacement therapy? Yes No |
| 7. | Please select what hormones you are taking and/or the name of your medication: |
| | Testosterone |
| | Estrogen |
| | Progesterone |
| | Thyroid |
| | Other: |
| 8. | Medication Name if known: |
| 9. | At what age did your periods begin? |
| 10 | D. Do you still have regular periods? Yes No |
| 13 | 1. If you answered No on question 10, please select one of the following reasons: |

| Melanoma | , Pancreatic, Stomach, Uter istory of cancer Family | • | |
|---|---|---|---|
| Melanoma No Family h Mother Father Sibling Grandmother Grandfather Aunt | , Pancreatic, Stomach, Uter istory of cancer Family | ine, Thyroid, Colon, and/or Sa<br>history unknown<br>mediate Family | |
| Melanoma No Family h Mother Father Sibling Grandmother Grandfather | , Pancreatic, Stomach, Uter istory of cancer Family | ine, Thyroid, Colon, and/or Sa<br>history unknown<br>mediate Family | |
| Melanoma No Family h Mother Father Sibling Grandmother | , Pancreatic, Stomach, Uter istory of cancer Family | ine, Thyroid, Colon, and/or Sa<br>history unknown<br>mediate Family | |
| Melanoma No Family h Mother Father Sibling | , Pancreatic, Stomach, Uter istory of cancer Family | ine, Thyroid, Colon, and/or Sa<br>history unknown<br>mediate Family | |
| Melanoma No Family h Mother Father | , Pancreatic, Stomach, Uter istory of cancer Family | ine, Thyroid, Colon, and/or Sa<br>history unknown<br>mediate Family | |
| Melanoma No Family h Mother Father | , Pancreatic, Stomach, Uter | ine, Thyroid, Colon, and/or Sa | |
| Melanoma No Family h | , Pancreatic, Stomach, Uter | ine, Thyroid, Colon, and/or Sa | |
| Melanoma<br>□No Family h | , Pancreatic, Stomach, Uter | ine, Thyroid, Colon, and/or Sa | |
| Melanoma | , Pancreatic, Stomach, Uter | ine, Thyroid, Colon, and/or Sa | |
| Melanoma | , Pancreatic, Stomach, Uter | ine, Thyroid, Colon, and/or Sa | |
| | | • | |
| | 17. Please list below, any members of your family that have or have had: Breast, Ovarian, Prostate, Melanoma, Pancreatic, Stomach, Uterine, Thyroid, Colon, and/or Sarcoma. | | |
| | | Surgery Radiation | No Further details: |
| | | Chemo | Yes |
| Cancer Type | Year of diagnosis | Treatment | Treatment ongoing |
| 16. In the char | t below please list any canc | , | |
| | aken any immune suppress<br>Yes Describe: | ant medication today? | |
| | aken any prescription anti-ir<br>Yes Describe: | nflammatory medication in the | e past 24 hours? |
| 13. Have you taken any over the counter anti-inflammatory medication in the past 8 hours? No Yes Describe: | | | |
| Section 3: In section 3 you will find questions about medications you may have taken today. | | | |
| 12. Do you stil<br>☐Both | I have one or both ovaries? One None | | |
| Other ( | please describe): | | |
| <u>=</u> | | | |
| Unknov | Ablation | | |
| Uterine Unknow | Response to Birth Control | | |
| Respor Uterine Unknow | ectomy<br>ise to Birth Control | | |
| Respor Uterine Unknow | ectomy | | |

| Jncle Cousin 18. What Proced | | | | | |
|---|---|---|---|---|---|
| Cousin 18. What Proced | | | | | |
| 18. What Proced | | | | | |
| ☐Screening Mammogram | | | | | |
| _ | _ | | | | |
| ☐ Diagnostic Mammogram | | | | | |
| ☐ Screening Ultrasound | | | | | |
| ☐ Diagnostic Ultrasound | | | | | |
| □Biopsy | | | | | |
| ☐Screening<br>— | | | | | |
| □Diagnostic | c MRI | | | | |
| □Other: | | | | | |
| □ottlei. — | | | | | |
| □otner | | | | | |
| | St | udy Participant | Stop H | lere | |
| | St | udy Participant | Stop H | lere | |
| | St<br>Collection Time | udy Participant | _ | lere Distance for | Distance for |
| | | | _ | | Distance for Sample B |
| Collection Date C | | | _ | Distance for | |
| Collection Date Collection | | | _ | Distance for | |
| | | | _ | Distance for | |
| Collection Date Collection | | | _ | Distance for | |
| Collection Date Collection | | | _ | Distance for | |
| Collection Date Collection Notes: | | | _ | Distance for | |
| Collection Date Collection | | | itials | Distance for | |

# **Tear Based Breast Cancer Detection Clinical Information**

| Sample ID: | Collection | date: | Collectio | n time: |
|---|---|---|---|---|
| Initials: | | | | |
| Age: | Patient Heigh | nt: | Patient Weigh | nt: |
| Fatty Scatte Hetero | lect Patient's Breast Density (<br>red Fibroglandular Densities<br>ogeneously Dense<br>nely Dense | Category: | | |
| 2. Has patie Yes No | ent had previous biopsies? | | | |
| 3. Has the p Yes No | patient had at least one biops | y with atypica | l hyperplasia? | |
| Screer Screer Screer Diagno | rocedures below, if conducted in ing Mammogram in ing Ultrasound in ing MRI in its interest of the interest of | d at your clinic Normal Normal Normal Normal Normal Normal Positive | Called back Docate Called back Docate Called Back Docate Back Doca | ate:<br>ate:<br>ate:<br>ate:<br>ate: |
| 5. BiRads So | core 2 3 4 5 | <u> </u> | | |
| ☐6 mon<br>☐6 mon<br>☐Returr | the following was recommenth follow up (not high risk) th follow up (high risk screenined to normal screening I Exam follow-up (patient to y | ng protocol) | | ning) |
| 7. Were cal | cifications identified? | | | |
| LCIS Atypic Atypic | received a biopsy with Atypical Ductal Hyperplasia al Lobular Hyperplasia (describe): | cal results ple | ase indicate type of a | ntypia: |

| 9. If Benign please select or describe: Hyperplasia of usual type Benign Calcifications Papilloma Sclerosing Adenosis Fat Epithelial Atypia Fibroadenoma Radial Scar Stromal Fibrosis Calcifications Fibrocystic Change | |
|---|---|
| 10. The following information is requested | for positive diagnosis: |
| Breast Cancer type and location | Receptors: |
| □DCIS □ left □right □ bila | teral ER+ |
| | teral ER- |
| | teral HER2 + |
| | teral HER2 – |
| | teral PR + |
| Other: | □PR- |
| 11. Metastasis: Yes:No | <u> </u> |
| 12. Tumor Grade | 13. Stage if known: |
| ∏gx | 0 |
| G1-low grade | ☐ la ☐ lb |
| G2-intermediate grade | ☐ IIa ☐ IIb |
| G3-high grade | ☐ IIIa ☐ IIIb ☐ IIIc |
| G4-high grade | ☐ Iva ☐ IVb |
| 14. Ki67 | 15. Tumor/s Size |
| ∐High | |
| Borderline | |
| Low | |